CLINICAL TRIAL: NCT01654601
Title: Clinical Trials to Compare the Pharmacokinetics Profile of DWCZP Tablet 100mg and Clozaril® Tablet 100mg After a Multi-dose Oral Administration in Schizophrenia Patients
Brief Title: A Study to Compare the Pharmacokinetics Profile of DWCZP Tablet 100mg and Clozaril® Tablet 100mg
Acronym: DWCZP-I-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong Wha Pharmaceutical Co. Ltd. (Industry)
Collaborators: The Catholic University of Korea (Other); Konkuk University Hospital (Other); Naju National Hospital (Other); Seoul National Hospital (Other Government); Wonkwang University (Other); DongGuk University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DWCZP-I-1
Record Dates: First submitted 2012-07-25; First posted 2012-08-01 (Estimated); Results first posted 2014-03-14 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Clozapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A Group (Experimental): 1.1st Administration - DWCZP tablet 100mg Mutiple dose
  2.2nd Administration - Clozaril tablet 100mg Mutiple dose
  Interventions: Drug: DWCZP; Drug: Clozaril
- B Group (Experimental): 1.1st Administration - Clozaril tablet 100mg Mutiple dose
  2.2nd Administration - DWCZP tablet 100mg Mutiple dose
  Interventions: Drug: DWCZP; Drug: Clozaril

INTERVENTIONS:
Drug: DWCZP — Multiple dose
  Other Names: DWCZP Tablet 100mg
Drug: Clozaril — multiple-dose
  Other Names: Clozaril Tablet 100mg

SUMMARY:
To evaluate the pharmacokinetics of oral multiple-dose of DWCZP tablet 100mg.

DETAILED DESCRIPTION:
A randomized, 2-way crossover, open, phase I study to compare the pharmacokinetics profile of DWCZP tablet 100mg and Clozaril® tablet 100mg after a multiple-dose oral administration in schizophrenia patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female within range of 20 to 60.
* Diagnosed as Schizophrenia (Note: Diagnosed with DSM-IV, ICD-10 as a standard Schizophrenia diagnostic tool).
* Administered clozapine for 3 months before signing agreement with same amount daily and who can administer clozapine 100mg twice (morning, evening) a day, total of 200mg during the study time.
* One who might be pregnant must get negative result for pregnancy test (urine or blood β-hCG) before the randomization and during the study time, one must agree appropriate contraception. However, one who is using only hormone-contraceptive for birth control and has not been more that 1 year after Tubal ligation or menopause are excluded.
* One who understood completed about this study after the explanation is given, decided to volunteer and gave written informed consent approved by IRB to participate in study in compliance with the requirement of the entire protocol.

Exclusion Criteria:

* One who has record of hypersensitive reaction with Clozapine or other antipsychotic drug.
* WBC count less than 4,000/ml or Absolute Neutrophil count less than 2,000/ml.
* Administering hypertension drug or has orthostatic hypotension.
* One who has clinical problem with kidney or liver and include following criteria: CCr < 50mL/min; BUN > 30 mg/dl; ALT 또는 AST > 3 x ULN; Total bilirubin > 2 x ULN; ALP > 2 x ULN.
* Diagnosed to have other psychiatric or neurological problems other than Schizophrenia (e.g., Organic mental disorder, severe tardive dyskinesia, idiopathic Parkinson's disease, etc).
* Record of Granulocytopenia or Myeloproliferative disorder in the past.
* Record of stomach-related problems(active Crohn's disease, vital infectious intestine disease, ulcer, acute or chronic pancreatitis etc) or surgery which can affect absorption of study drug. However, simple appendectomy or herniotomy are exceptions.
* Chronic Hepatitis B carrier, proof of Hepatitis C carrier or Hepatitis C antibody.
* Immunodeficiency diseases such as HIV positive, AIDS, had bone marrow transplantation or has blood ammonia.
* Record of seizure in 1 year before signing informed consent form or had administered anti-seizure drug before(e.g., Epilepsy, Convulsions, Myasthenia gravis, etc).
* One who constantly drinks(> 21Units/week, 1Unit = 10g of pure alcohol) or cannot stop drinking alcohol during hospitalization period.
* Smoking past 3 months before signing informed consent form or cannot stop smoking during hospitalization period.
* One who cannot attend routine blood tests.
* Bone marrow malfunction.
* Mental illness, durg addicted or in coma.
* One who has any kind of circulation imperfection and patient with depressed central nervous system.
* Major kidney and heart problem(e.g. myocarditis).
* Incurable epilepsy.
* Paralytic intestinal obstruction.
* Generic problems such as Lactose intolerance, Galactose intolerance, Lapp lactose deficiency, Glucose-Galactose absorption deficiency, etc.
* Administered barbital-related drugs and drug metabolizing enzyme inducer and inhibitor in 1 month before starting the study.
* One who had drugs that can affect on result of the study for past 10 days before the study start.
* One who had whole blood donation in 2 months or blood component donation or transfusion in 1 month before signing the informed consent form.
* Attended clinical tests or bioequivalence tests in 2 months before signing informed consent form.
* Currently pregnant or breast-feeding or has possibility of pregnancy because one is not using medically approved contraception(Note: condoms, oral contraceptive, intrauterine device, abstinence etc).
* One who is clinically significant by observations considered as unsuitable based on medical judgement by investigators.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2012-06; Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Won-Myoung Bahk, M.D., Principal Investigator — The Catholic University of Korea, Yeouido St.Mary's Hospital
Locations (5):
- South Korea (5):
  - Konkuk University Hospital, Choongju
  - Wonkwang University, Iksan
  - Naju National Hospital, Naju
  - The Catholic University of Korea, yeouido St.Mary's Hospital, Seoul
  - Seoul National Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Catholic University of Korea, Yeouido St.Mary's Hospital — http://www.cmcsungmo.or.kr/
- See also: Konkuk University Hospital — http://www.kuh.co.kr
- See also: Naju National Hospital — http://www.najumh.go.kr
- See also: Seoul National Hospital — http://www.ncmh.go.kr
- See also: Wonkwang University — http://www.wkuh.org/
- See also: Dongguk University — http://www.dumc.or.kr

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from a specialty clinic at s hospital, in Seoul, Naju, Chungju, Iksan and Kyungju, Korea between June 2012 and March 2013
Pre-assignment Details: 32 participantsrecruited : 28 screened, 4 excluded(3 did not meet inclusion criteria and 1 refused participation)
Groups:
- A Group: DWCZP tablet 100mg twice daily in first intervention period and Clozaril tablet 100mg twice daily in second intervention period (no washout period, Intervention period : 10days)
- B Group: Clozaril tablet 100mg twice daily in first intervention period and DWCZP tablet 100mg twice daily in second intervention period (no washout period, Intervention period : 10days)
Period: 1st Administration
Arm/Group | A Group | B Group
Started | 14 | 14
Completed | 12 | 12
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Protocol Violation | 0 | 2
Period: 2nd Administration
Arm/Group | A Group | B Group
Started | 12 | 12
Completed | 11 | 11
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A Group | B Group | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 6 | 8 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 14 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration of Clozapine in Plasma
Time Frame: Up to 12hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | A Group | B Group
Number analyzed (Participants) | 11 | 11
ng/mL | 524.62 (272.51) | 551.18 (263.26)

2. Secondary Outcome: Time to Reach Maximum Concentration of Clozapine in Plasma
Time Frame: Up to 12hours
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | A Group | B Group
Number analyzed (Participants) | 11 | 11
hour | 2.43 (1.71) | 2.75 (1.93)

3. Secondary Outcome: Terminal Half Life of Clozapine in Plasma
Time Frame: Up to 12hours
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | A Group | B Group
Number analyzed (Participants) | 11 | 11
hour | 11.98 (6.89) | 10.88 (3.81)

4. Secondary Outcome: Accumulation Rate of Clozapine in Plasma
Time Frame: Up tp 12hours
Measure: Mean (Standard Deviation); unit: ng/ml/hr
Arm/Group | A Group | B Group
Number analyzed (Participants) | 11 | 11
ng/ml/hr | 2.01 (0.81) | 1.88 (0.44)

ADVERSE EVENTS:
Time Frame: 3 weeks
Description: abnormal vital sign, physical examination, electrocardiogram or laboratory finding after study drug adminstration
Arm/Group | A Group | B Group
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/14
Other Adverse Events (participants affected / at risk) | 5/14 | 4/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A Group (N=14) | B Group (N=14)
Fracture of distal clavicle, Lt. (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A Group (N=14) | B Group (N=14)
Nausea (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Ocular discomfort (Eye disorders) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Apathy (Psychiatric disorders) | 1 | 0
Dysmenorthoea (Reproductive system and breast disorders) | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No